CLINICAL TRIAL: NCT03260517
Title: A Clinical PeRformance EVAluatIon of a New Medtronic Coronary Drug-Coated BaLloon Catheter for the Treatment of De Novo Lesions, In-Stent Restenosis and Small Vessel Disease in Coronary Arteries: The PREVAIL Study
Brief Title: The PREVAIL Study
Acronym: PREVAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17027DCB001
Record Dates: First submitted 2017-08-10; First posted 2017-08-24 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: In-stent Restenosis; Ischemic Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Mdt Drug-Coated Balloon) (Experimental): Medtronic Coronary Drug-Coated Balloon Catheter used for dilatation of the target lesion.
  Interventions: Device: Medtronic Coronary Drug-Coated Balloon Catheter

INTERVENTIONS:
Device: Medtronic Coronary Drug-Coated Balloon Catheter — Medtronic Paclitaxel Coronary Drug-Coated Balloon Percutaneous transluminal coronary angioplasty

SUMMARY:
To evaluate the clinical safety and efficacy of a new Medtronic Coronary Drug-Coated Balloon Catheter in the treatment of de novo lesions, small vessel disease or In-Stent Restenosis with coronary lesions previously treated with drug-eluting or bare metal stents in native coronary arteries.

DETAILED DESCRIPTION:
This study is a prospective, pre-market, multi-center, single arm study evaluating up to 50 subjects with symptoms of ischemic heart disease attributable to stenotic lesions of the coronary arteries that are amenable to treatment with the Medtronic Coronary Drug-Coated Balloon Catheter.

Patients with de novo lesions, In-Stent Restenosis or small vessel disease who qualify for percutaneous coronary interventions treatable with the device with a diameter between 2.0 mm to 4.0 mm and a length ≤25 mm will be screened and are intended to participate in this study.

Each subject is expected to be followed in the study for 12 months. Procedural/acute outcomes and clinical outcomes will be assessed at procedure, 30 days, 6 and 12 months.

ELIGIBILITY:
Key Inclusion Criteria

* Subject with documented stable or unstable angina, and/or clinical evidence of ischemia
* Subject is an acceptable candidate for treatment with a Coronary Drug- Coated Balloon in accordance with the applicable guidelines on percutaneous coronary interventions, manufacturer's Instructions for Use and the Declaration of Helsinki.

Key Exclusion Criteria

* Acute Myocardial Infarction within the previous 72 hours
* Planned treatment involves a bifurcation
* Three vessel disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
In-stent (in balloon) Late Lumen Loss (LLL) as measured by Quantitative coronary angiography (QCA) at six months | At 6 months follow up
  The average 6 months in-stent (in-balloon) LLL will be compared to a maximum acceptance rate. If in-stent (in-balloon) LLL is less than the maximum acceptance rate, then the trial will be considered to have met the primary endpoint.

SECONDARY OUTCOMES:
All deaths including cardiac death.procedure | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedure
Target Vessel Myocardial Infarction (TVMI) | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedure
Major adverse cardiac event (MACE) defined as composite of death, Myocardial infarction (MI), emergent Coronary Artery Bypass Graft (CABG) or repeat Target lesion revascularization (TLR) (clinically driven) by percutaneous or surgical methods | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedures
Target vessel failure (TVF) defined as cardiac death, TVMI, or clinically-driven Target vessel revascularization (TVR) by percutaneous or surgical methods. | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedures
5. Target lesion failure (TLF) defined by a composite of cardiac death, TVMI, or clinically-driven TLR by percutaneous or surgical methods. | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedure
All revascularizations (TLR, TVR and non-TVR). | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedure
Stent Thrombosis rate as defined as definite, probable, possible, and overall stent thrombosis (according to Academic Research Consortium definition). | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedure
Acute success (device, lesion and procedure success). | 30 days, 6 months and 1 year after procedure
  Clinical endpoints to be assessed at 30 days, 6 months and 1 year after procedure

OTHER OUTCOMES:
In-stent (balloon) and in-segment LLL | 6 months post-procedure
  Angiographic Endpoints to be assessed at 6 months post-procedure
In-stent (balloon) and in-segment percent diameter stenosis (%DS (Percent diameter stenosis)). | 6 months post-procedure
  Angiographic Endpoints to be assessed at 6 months post-procedure
In-stent (balloon) and in-segment Binary Angiographic Restenosis (BAR) rate [defined as ≥50% diameter stenosis (DS)]. | 6 months post-procedure
  Angiographic Endpoints to be assessed at 6 months post-procedure
In-stent (balloon) and in-segment Minimum luminal/lumen diameter (MLD). | 6 months post-procedure
  Angiographic Endpoints to be assessed at 6 months post-procedure

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - CHU Liege, Liège
- Italy (2):
  - IRCCS Policlinico San Donato, Milan
  - Ospedale San Raffaele, Milan
- Netherlands (5):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - Haga Ziekenhuis locatie Leyweg, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grosso A, Neves de Faria RI, Bojke L, Donohue C, Fraser CI, Harron KL, Oddie SJ, Gilbert R. Cost-effectiveness of strategies preventing late-onset infection in preterm infants. Arch Dis Child. 2020 May;105(5):452-457. doi: 10.1136/archdischild-2019-317640. Epub 2019 Dec 13. PMID 31836635